CLINICAL TRIAL: NCT06468098
Title: Phase Ib Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of IBI363 Combination Therapy in Subjects With Advanced Malignancies
Brief Title: A Study of IBI363 in Subjects With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363A103
Record Dates: First submitted 2024-06-13; First posted 2024-06-21 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): IBI363 combined with chemotherapy in patients with advanced NSCLC who have failed at least one prior line of standard therapy (which needs to include immunotherapy)
  Interventions: Drug: IBI363 + chemotherapy
- Cohort 2A (Experimental): IBI363 combined with chemotherapy as first-line in patients with advanced colorectal cancer, including a safety run-in phase and a randomized controlled phase
  Interventions: Drug: IBI363 + chemotherapy
- Cohort 2B (Experimental): IBI363 combined with chemotherapy as first-line in patients with advanced colorectal cancer, including a safety run-in phase and a randomized controlled phase
  Interventions: Drug: IBI363 + chemotherapy
- Cohort 3 (Experimental): IBI363 combined with chemotherapy in patients with advanced biliary tract tumors that have failed or are intolerant to first-line standard therapy
  Interventions: Drug: IBI363 + chemotherapy
- Cohort 4 (Experimental): IBI363 combined with chemotherapy in second-line in patients with Advanced Esophageal Squamous Cell Carcinoma
  Interventions: Drug: IBI363 + chemotherapy
- Cohort 5 (Experimental): IBI363 combined with chemotherapy in second-line in patients with Advanced Gastric Cancer
  Interventions: Drug: IBI363 + chemotherapy
- Cohort 6 (Experimental): IBI363 combined with chemotherapy in patients with Advanced Triple-Negative Breast Cancer
  Interventions: Drug: IBI363 + chemotherapy
- Cohort 7 (Experimental): IBI363 combined with chemotherapy in patients with platinum-resistant ovarian cancer that has failed or is intolerant to standard therapy
  Interventions: Drug: IBI363 + chemotherapy
- Cohort 8 (Experimental): IBI363 Combined with Investigator's Choice Standard of Care(SOC) in Patients with Advanced Solid Tumors
  Interventions: Drug: IBI363 + Investigator's Choice SOC

INTERVENTIONS:
Drug: IBI363 + chemotherapy — In this group, patients will receive IBI363 and chemotherapy
  Arms: Cohort 1; Cohort 2A; Cohort 2B; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7
Drug: IBI363 + Investigator's Choice SOC — In this group, patients will receive IBI363 and Investigator's Choice SOC
  Arms: Cohort 8

SUMMARY:
This is an open-label, multicenter Phase Ib study to evaluate the safety, tolerability, and efficacy of IBI363 in advanced malignancies patients

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent and be able to comply with the program's visit schedule and related procedures.
2. Male or female subjects, age 18~75 years.
3. Histologically or cytologically confirmed advanced malignancy.
4. Subjects who have progressed on standard therapy, who are unsuitable for standard therapy, who do not have standard therapy, or who have refused standard therapy. For particular cohort, subjects who have not received prior systemic therapy for advanced disease.
5. At least one measurable lesion (target lesion) per RECIST v1.1.
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
7. Life expectancy of 3 months or more.
8. Female subjects of childbearing age or male subjects whose partners are female subjects of childbearing age agree to strictly adopt effective contraceptive measures throughout the entire treatment period and 6 months after the treatment period.

Exclusion Criteria:

1. Women who are pregnant or lactating, or intending to become pregnant before, during, or within 6 months after the last dose of study drug.
2. Active or untreated CNS metastases confirmed by imaging evaluation during screening or previous imaging evaluation. Patients with asymptomatic brain metastases may participate in this study.
3. History of active thrombosis or deep vein thrombosis or pulmonary embolism within 4 weeks prior to the first dose of study drug.
4. Clinically significant cardiovascular or cerebrovascular disease.
5. Interstitial pneumonia, pulmonary fibrosis, pneumoconiosis, drug-associated pneumonia, and radiation pneumonitis requiring steroid hormone or other therapy, as well as history of severe abnormal lung function or other forms of restrictive lung disease.
6. History of allergies, asthma, atopic dermatitis.
7. Concomitant pleural or pericardial effusion requiring repeated drainage or with significant symptoms.
8. Active autoimmune disease requiring systemic therapy within 2 years prior to first dose.
9. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
10. Subjects with known or suspected hypersensitivity to the study drug and any excipients.
11. Subject has a prior history of significant toxicity associated with immune checkpoint inhibitor administration that requires permanent discontinuation.
12. Subjects with unresolved > Grade 1 toxicity associated with any prior antineoplastic therapy, with the exception of persistent Grade 2 alopecia, peripheral neuropathy, hypomagnesemia, and toxicities that are not expected to be reversible but are stably controlled by medications (e.g., hypothyroidism stably controlled by substitution therapy, hypertension stably controlled by antihypertensive medications with a BP of less than 160/100 mmHg).
13. Inadequate recovery from previous surgery or any major surgery within 4 weeks prior to the first dose of study drug.
14. Active uncontrolled bleeding or known bleeding tendency.
15. Subject has a current or recent (within 6 months) major gastrointestinal disease or condition.
16. Subjects with uncontrolled tumor-related pain or symptomatic hypercalcemia.
17. Known positive HIV test, active hepatitis B, hepatitis C (HCV), tuberculosis.
18. Severe/active/uncontrolled infection, infection requiring systemic intravenous antibiotic therapy, or unexplained fever within 2 weeks prior to the first dose of study drug.
19. Diagnosis of another malignancy within 5 years prior to the first dose, exceptions include radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radically resected carcinoma in situ, as well as post-radical localized prostate cancer, and papillary thyroid cancer.
20. Exclusion of contraindications to combination medications including, but not limited to: known contraindications to irinotecan therapy for the combination irinotecan or liposomal irinotecan cohort including, but not limited to: having the UGTA1*6/*6, UGT1A1*28/*28, or UGT1A1*6/*28 genotypes; history of prior pelvic and abdominal radiotherapy.
21. Presence of any disease, treatment or laboratory test abnormality, or history or current evidence of substance abuse that, in the judgment of the investigator, may compromise the safety of the subject, interfere with obtaining informed consent, affect subject compliance, or compromise the safety evaluation of the study drug.
22. Mental illness, presence of altered mental status, or substance abuse that prevents understanding of the informed consent process and/or completion of necessary study-related evaluations.
23. For known or foreseeable reasons, the Investigator believes that the subject is unable to fulfill the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Enent (AE) | Up to 90 days after the last administration
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0
Treatment-Emergent AE (TEAE) | Up to 90 days after the last administration
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0
Adverse Event of Special Interest (AESI) | Up to 90 days after the last administration
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0
Serious Adverse Event (SAE) | Up to 90 days after the last administration
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0
Objective response rate (ORR) | Through out the study (up to 2 years)
  ORR is defined as the proportion of participants with a complete response (CR) or partial response (PR).
disease control rate (DCR) | Through out the study (up to 2 years)
  DCR is defined as the proportion of participants with a complete response (CR) or partial response (PR) or stable disease(SD)
time to response (TTR) | Through out the study (up to 2 years)
  TTR is defined as the time from the date of first dose of study drug to the date of first documented tumor response (CR/PR)
duration of response (DoR) | Through out the study (up to 2 years)
  DoR is defined as the time from the date of first documented tumor response (CR/PR) until PD/death
progression-free survival (PFS) | Through out the study (up to 2 years)
  PFS is defined as the time from the date of first dose of study drug to the date of the first documented progression or death due to any cause, whichever occurs first
Overall survival (OS) | Through out the study (an average of 2 years)
  OS is defined as the time from the date of first dose of study drug until the date of death from any cause.

SECONDARY OUTCOMES:
Plasma concentration (Cmax) of IBI363 | Up to 2 years
  PK parameters maximum concentration (Cmax) of IBI363
Area under the curve (AUC) of IBI363 | Up to 2 years
  PK parameters area under the curve (AUC)?of IBI363
Half-life (T1/2) of IBI363 | Up to 2 years
  PK parameters half-life (t1/2)?of IBI363
Clearance (CL) of IBI363 | Up to 2 years
  PK parameters clearance rate of IBI363
Volume of distribution (V) of IBI363 | Up to 2 years
  PK parameters apparent volume of distribution(V)?of IBI363
Immunogenicity of IBI363 | Up to 2 years
  Incidence of anti-drug (IBI363) antibody

CONTACTS AND LOCATIONS:
Overall Officials: tingbo Liang, M.D., Principal Investigator — The First Affiliated Hospital ZJ University; xueli Bai, M.D., Principal Investigator — The First Affiliated Hospital ZJ University; jianming Xu, M.D., Principal Investigator — Chinese PLA General Hospital; shun Lu, M.D., Principal Investigator — Shanghai Chest Hospita; tao Zhang, M.D., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Shanghai Chest Hospita, Shanghai, Shanghai Municipality, China